CLINICAL TRIAL: NCT01910610
Title: Multi-Line Therapy Trial in Unresectable Wild-Type RAS Metastatic Colorectal Cancer. A GERCOR Randomized Open-label Phase III Study.
Brief Title: Multi-Line Therapy Trial in Unresectable Metastatic Colorectal Cancer
Acronym: STRATEGIC-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STRATEGIC-1 C12- 2; 2013-001928-19 (EudraCT Number)
Record Dates: First submitted 2013-07-23; First posted 2013-07-29 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer Metastatic
Keywords: wild-type RAS metastatic colorectal cancer
MeSH Terms: interventions — Bevacizumab; Panitumumab; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STRATEGY A (Experimental): FOLFIRI-cetuximab, followed by oxaliplatin-based chemotherapy with bevacizumab
  Interventions: Biological: FOLFIRI-cetuximab; Biological: mFOLFOX6-bevacizumab; Biological: XELOX + bevacizumab
- STRATEGY B (Experimental): OPTIMOX-bevacizumab, followed by irinotecan-based chemotherapy with bevacizumab, followed by anti-EGFR mab with or without irinotecan
  Interventions: Biological: OPTIMOX-bevacizumab; Biological: irinotecan-based chemo + bevacizumab; Biological: Anti-EGFR agent (cetuximab +/- irinotecan or panitumumab); Biological: XELOX + bevacizumab

INTERVENTIONS:
Biological: FOLFIRI-cetuximab
  Arms: STRATEGY A
Biological: mFOLFOX6-bevacizumab
  Arms: STRATEGY A
Biological: OPTIMOX-bevacizumab
  Arms: STRATEGY B
Biological: irinotecan-based chemo + bevacizumab
  Arms: STRATEGY B
Biological: Anti-EGFR agent (cetuximab +/- irinotecan or panitumumab)
  Arms: STRATEGY B
Biological: XELOX + bevacizumab

SUMMARY:
STRATEGIC-1 is a study designed to determine the best sequence of therapy in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
This is a phase III study assessing 2 mutli-line therapeutic strategies in patients with unresectable wild-type RAS metastatic colorectal cancer. All the available treatments are being used in each strategy (oxaliplatine, irinotecan, fluoropyrimidines, bevacizumab, cetuximab or panitumumab) but in a different order:

STRATEGY A: FOLFIRI-cetuximab, followed by oxaliplatin-based chemotherapy with bevacizumab vs.

STRATEGY B: OPTIMOX-bevacizumab, followed by irinotecan-based chemotherapy with bevacizumab, followed by anti-EGFR mab with or without irinotecan.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent, and willing and able to comply with protocol requirements,
2. Histologically proven adenocarcinoma of the colon and/or rectum,
3. Wild-type RAS tumor no mutation in exon 2 [codon 12/13], exon 3 [codon 59/61] and exon 4 [codon 117/146] of both KRAS and NRAS genes (local assessment, performed either on primary tumor or metastasis), In exceptional circumstances, RAS mutational status (KRAS and NRAS) can be pending at time of randomization, provided it is obtained within the first two cycles of first line therapy
4. Metastatic disease confirmed,
5. No prior therapy for metastatic disease (in case of previous adjuvant therapy, interval from end of chemotherapy and relapse must be >6 months for fluoropyrimidine alone or >12 months for oxaliplatin-based, bevacizumab-based, or cetuximab-based therapy),
6. Duly documented unresectable metastatic disease, ie not suitable for complete carcinological surgical resection at inclusion [NB: patients with unresectable disease at study entry but with any potential of salvage surgery after induction therapy are eligible],
7. At least one measurable or evaluable lesion as assessed by CT-scan or MRI (Magnetic Resonance Imaging) according to RECIST v1.1,
8. Age ≥18 years,
9. ECOG Performance status (PS) 0-2,
10. Hematological status: neutrophils (ANC) ≥1.5x109/L; platelets ≥100x109/L; haemoglobin ≥9g/dL,
11. Adequate renal function: serum creatinine level <150µM,
12. Adequate liver function: serum bilirubin ≤1.5 x upper normal limit (ULN), alkaline phosphatase <5xULN,
13. Proteinuria <2+ (dipstick urinalysis) or ≤1g/24hour,
14. Baseline evaluations performed before randomization when the KRAS WT status is known: clinical and blood evaluations no more than 2 weeks (14 days) prior to randomization, tumor assessment (CT-scan or MRI, evaluation of non-measurable lesions) no more than 3 weeks (21 days) prior to randomization,
15. Female patients must commit to using reliable and appropriate methods of contraception during the trial and until at least six months after the end of study treatment (when applicable). Male patients with a partner of childbearing potential must agree to use contraception in addition to having their partner use another contraceptive method during the trial and until at least 6 months after the end of the study treatment,
16. Registration in a national health care system (CMU included for France).

Exclusion Criteria:

1. History or evidence upon physical examination of CNS metastasis (e.g. non irradiated CNS metastasis, seizure not controlled with standard medical therapy), unless adequately treated,
2. Exclusive bone metastasis,
3. Uncontrolled hypercalcemia,
4. Pre-existing permanent neuropathy (NCI grade ≥2),
5. Uncontrolled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg), or history of hypertensive crisis, or hypertensive encephalopathy,
6. Concomitant unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy),
7. Treatment with any investigational medicinal product within 28 days prior to study entry,
8. Other serious and uncontrolled non-malignant disease,
9. Gilbert's syndrome,
10. Other concomitant or previous malignancy, except: i/ adequately treated in-situ carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for >5 years,
11. Major surgery (open biopsy, surgical resection, wound revision or any other major surgery involving entry into body cavity) or significant traumatic injury within the last 28 days prior to randomization, and/or minor surgical procedure including placement of a vascular device within 2 days of first study treatment,
12. Pregnant or breastfeeding women,
13. Patients with known allergy/hypersensitivity to any component of study drugs,
14. History of arterial thrombo and/or embolic event (e.g. myocardial infarction, stroke,…) within 6 months prior to randomization,
15. Chronic inflammatory bowel disease
16. Total bowel obstruction,
17. History of abdominal fistula, GI perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to randomization,
18. Serious, non-healing wound, active ulcer or untreated bone fracture,
19. History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding,
20. Current or recent (within 10 days of randomization) use of aspirin (>325 mg/d), clopidogrel (>75 mg/d) or use of oral anticoagulants or thrombolytic agents.
21. Concomitant administration of live, attenuated virus vaccine such as yellow fever vaccine
22. Concomitant administration of prophylactic phenytoin.
23. Treatment with sorivudine or its chemically related analogues, such as brivudine.
24. Patients with known dihydropyrimidine dehydrogenase (DPD) deficiency.
25. Concomitant use with St John's Wort
26. Patients with interstitial pneumonitis or pulmonary fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Duration of Disease Control (DDC) | From baseline until end of strategy; up to 80 months after the beginning of the study
  DDC is defined as the sum of PFS of each active treatment course planned in the treatment strategy. DDC excludes 1) intervals between disease progression and re-initiation of treatment, and 2) PFS of inactive treatment if PD occurs at first evaluation after treatment re-initiation (either reintroduction in a stop-and-go strategy or subsequent course of treatment in a multi-line strategy).

SECONDARY OUTCOMES:
Assessment of Quality of life (QoL) | From baseline until end of strategy; up to 80 months after the beginning of the study
  QoL will be considered to be improved if at least one time to QoL score deterioration (5 targeted dimensions) will be significantly longer without a significant shorter time to QoL score dimensions for other 4 targeted dimensions.
Overall Survival (OS) | Up to 80 months after the beginning of the study
  Time from randomization to the date of death from any cause
Time to Failure of Strategy (TFS) | Up to 80 months after the beginning of the study
  TFS is defined as beginning with the initiation of the strategy under investigation and ending with the first of the following events: 1) death, 2) disease progression on the last received planned sequence, 3) patient requires the addition of a new (unplanned) therapeutic agent, 4) patient experiences disease progression during a partial or complete break in therapy from initial treatment strategy and receives no further therapy within one month.
Progression-free survival (PFS) per sequence of therapy | Up to 80 months after the beginning of the study
  Time from randomization to the date of first documented disease progression or death from any cause, whichever occurs first.
Tumor Response Rate (RR) | From baseline until end of strategy; up to 80 months after the beginning of the study
  Tumor response will be assessed using RECIST version 1.1 per sequence of therapy
Curative salvage surgery rate | From baseline until end of strategy; up to 80 months after the beginning of the study
  The number of patient with R0 and R1 curative salvage surgery will be assessed globally (per arm) and per sequence of therapy
Safety profile of each treatment sequence | From study entry to 1 month after last study drug administration; up to 80 months after the beginning of the study
  The report will take into account all adverse events observed during and after drug administration, including any adverse events that may be related to the administration procedure itself.

CONTACTS AND LOCATIONS:
Overall Officials: Benoist Chibaudel, MD, Principal Investigator — Institut Hospitalier Franco-Britannique
Locations (56):
- France (44):
  - Centre Hospitalier Annecy Gennevois, Annecy
  - Centre hospitalier Auxerre, Auxerre
  - Centre François Baclesse, Caen
  - Centre Hospitalier, Cannes
  - Centre Hospitalier Chateauroux, Châteauroux
  - Hospices Civils de Colmar, Colmar
  - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier, Dax
  - Centre d'oncologie et de radiothérapie du Parc, Dijon
  - Centre Georges François Leclerc, Dijon
  - CHD Vendée, La Roche-sur-Yon
  - Hôpital Louis Pasteur, Le Coudray
  - Hôpital Privé de l'Estuaire, Le Havre
  - Clinique Victor Hugo, Le Mans
  - Institut d'oncoloige Hartmann, Levallois-Perret
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Centre Bourgogne, Lille
  - Centre Hospitalier de Bretagne Sud, Lorient
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital Européen, Marseille
  - Hôpital Nord, Marseille
  - Centre Hospitalier Layné, Mont-de-Marsan
  - Centre d'oncologie de Gentilly, Nancy
  - Centre Sainte Catherine de Sienne, Nantes
  - Hôpital Cochin, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital Saint-Joseph, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Tenon, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Périgueux, Périgueux
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Clinique de l'Alliance, Saint-Cyr-sur-Loire
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - CH de Senlis, Senlis
  - Centre Hospitalier de Sens, Sens
  - Hôpital Broussais - CH Saint Malo, St-Malo
  - Clinique Sainte-Anne, Strasbourg
  - Hôpital Foch, Suresnes
  - Hôpitaux du Léman, Thonon-les-Bains
  - Hôpital Sainte Musse, Toulon
  - Clinique Générale, Valence
  - Institut de Cancérologie, Villeneuve-d'Ascq
- Ireland (10):
  - Bon Secours Hospital, Cork
  - Cork University Hospital, Cork
  - Adelaide & Meath Hospital Dublin ( AMNCH), Dublin
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - St. James's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Waterford, Waterford
- Israel (2):
  - Sheba Tel Hashomer, Ramat Gan
  - Assaf Harofeh Medical Center, Ẕerifin

REFERENCES:
- [Derived] Chibaudel B, Bonnetain F, Tournigand C, de Larauze MH, de Gramont A, Laurent-Puig P, Paget J, Hadengue A, Notelet D, Benetkiewicz M, Andre T, de Gramont A. STRATEGIC-1: A multiple-lines, randomized, open-label GERCOR phase III study in patients with unresectable wild-type RAS metastatic colorectal cancer. BMC Cancer. 2015 Jul 4;15:496. doi: 10.1186/s12885-015-1503-7. PMID 26141683